CLINICAL TRIAL: NCT04485130
Title: DISulfiram for COvid-19 (DISCO) Trial: A Phase 2 Double-Blind, Randomized Placebo-Controlled Trial of Disulfiram Compared to Standard Care in Patients With Symptomatic COVID-19
Brief Title: DISulfiram for COvid-19 (DISCO) Trial
Acronym: DISCO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low COVID case numbers, competing COVID treatments available
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Sulggi A. Lee, MD, PhD, Associate Professor of Medicine, University of California, San Francisco
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSF151837
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Covid19
Keywords: Disulfiram; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Disulfiram

STUDY DESIGN:
Intervention Model Description: This is a dose escalation double blind randomized (2:1) placebo-controlled trial of disulfiram given as 1000 mg/day x 5 consecutive days (Cohort 1: N=20 drug/N=10 placebo) or 2000 mg/day x 5 consecutive days (Cohort 2: N=20 drug/N=10 placebo) among 60 acute symptomatic lab-confirmed (<7 days) COVID+ individuals .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Disulfiram (Experimental): This study will provide disulfiram. Participants in Cohort 1 receiving disulfiram will take 2 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days. Participants in Cohort 2 receiving placebo will take 4 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
  Interventions: Drug: Disulfiram
- Placebo (Placebo Comparator): This study will provide placebo comparator for disulfiram. Participants in Cohort 1 receiving placebo will take 2 capsules of placebo (each capsule contains only microcrystalline cellulose powder) per day for a total of 5 consecutive days. Participants in Cohort 2 receiving placebo will take 4 capsules of placebo (each capsule contains only microcrystalline cellulose powder) per day for a total of 5 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Disulfiram — This study will provide disulfiram. Participants in Cohort 1 receiving disulfiram will take 2 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days. Participants in Cohort 2 receiving placebo will take 4 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
  Other Names: Antabuse
  Arms: Disulfiram
Drug: Placebo — This study will provide placebo. Participants in Cohort 1 receiving placebo will take 2 capsules of placebo (each capsule contains only microcrystalline cellulose powder) per day for a total of 5 consecutive days. Participants in Cohort 2 receiving placebo will take 4 capsules of placebo (each capsule contains only microcrystalline cellulose powder) per day for a total of 5 consecutive days
  Arms: Placebo

SUMMARY:
Disulfiram (DSF) a safe, easily dosed, FDA-approved drug for the treatment of alcohol dependence has been identified to be a potential therapeutic target for SARS-CoV-2 infection. Disulfiram may have both antiviral (inhibiting viral replication via blocking the Mpro protease and zinc ejection) and anti-inflammatory effects (via inhibition of NF-kB-induced and NLRP inflammasome-induced cytokine release) on SARS-CoV-2. We will study oral disulfiram given for 5 consecutive days (1000 mg/day in cohort 1; 2000 mg/day in cohort 2) in 60 symptomatic COVID+ individuals in a randomized (2:1) randomized, double blind placebo-controlled trial evaluating disulfiram's effect on COVID-19 symptom severity, SARS-CoV-2 viral load, and biomarkers of inflammation and pyroptosis (aberrant pro-inflammatory cell death) over 31 days.

DETAILED DESCRIPTION:
The identification of a safe, effective treatment for individuals with early mild-to-moderate symptomatic COVID-19 that prevent progression to more severe disease would have immediate public health implications. A hallmark of severe COVID-19 disease is immune system dysregulation called cytokine storm. Multiple studies have reported that patients with severe disease demonstrate elevated levels of pro-inflammatory cytokines early in disease, and elevated IL-6 plasma concentrations are predictive of poor clinical outcomes in COVID-19. Disulfiram, an FDA-approved drug for the treatment of alcohol dependence disorder is an appealing therapeutic option for COVID-19. It has a good safety profile, easy dosing schedule, and recent data suggesting multiple mechanisms by which disulfiram may act on COVID-19 (both as a direct antiviral agent as well as indirect effects on reducing inflammation). In addition disulfiram has been studied extensively with detailed available pharmacokinetic data; disulfiram has a short half-life ~7.5 hours with >90% of drug eliminated within 3 days post-dose, allowing quick reversal of any potential adverse effects. We will perform a phase 2 randomized (2:1), double blind placebo-controlled assessment of disulfiram in people with early mild-to-moderate symptomatic COVID-19. A total of 60 symptomatic COVID+ individuals will enrolled to receive active drug versus placebo (with equal distribution of mild or moderate/severe within each dosing cohort and within each randomization arm). For cohort 1, N=20 will receive DSF 1000 mg/N=10 placebo, and for cohort 2, N=20 will receive DSF 2000 mg/N=10 placebo. Drug/placebo will be administered using strict infection control protocols designed to support the study of people with acute COVID-19 infection per the Center for Diseases Control (CDC) guidelines (https://www.cdc.gov/coronavirus/2019-ncov/hcp/disposition-in-home-patients.html).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent, and
* Age >= 18 years, and
* SARS-CoV-2 positive PCR (nucleic acid) test within the preceding 7 days, and
* Not currently hospitalized, and
* Willing to abstain from any alcohol during the two week period in which disulfiram will be administered and during the two week period immediately after disulfiram administration.
* Both male and female subjects are eligible. Females of childbearing potential must have a negative pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Active malignancy requiring systemic chemotherapy or surgery in the preceding 3 months or for whom such therapies are expected in the subsequent 6 months
* Decompensated liver disease as defined by the presence of ascites, encephalopathy, esophageal or gastric varices, or persistent jaundice
* Serious illness requiring systemic treatment and/or hospitalization in the 3 months prior to study enrollment
* Concurrent treatment with immunomodulatory drugs, and/or exposure to any immunomodulatory drug in the 4 weeks prior to study enrollment (e.g. corticosteroid therapy equal to or exceeding a dose of 15 mg/day of prednisone for more than 10 days, IL-2, interferon-alpha, methotrexate, cancer chemotherapy). NOTE: use of inhaled or nasal steroid is not exclusionary.
* Serious medical or psychiatric illness that, in the opinion of the site investigator, would interfere with the ability to adhere to study requirements or to give informed consent.
* Current alcohol use disorder or hazardous alcohol use (>7 drinks per week for women or > 14 drinks per week for men) as determined by clinical evaluation.
* Current use of any drug formulation that contains alcohol or that might contain alcohol
* Current use of warfarin.
* Clinically active hepatitis determined by the study physician; ALT or AST > 3 x the upper limit of normal or total bilirubin outside the normal range.
* Allergy to rubber or thiuram derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sulggi A Lee, MD PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, Fresno, Fresno, California
  - San Francisco General Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
Planned sharing of de-identified individual participant data for the purposes of collaboration and meta-analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of study results
Access Criteria: De-identified data

REFERENCES:
- [Background] Lee SA, Elliott JH, McMahon J, Hartogenesis W, Bumpus NN, Lifson JD, Gorelick RJ, Bacchetti P, Deeks SG, Lewin SR, Savic RM. Population Pharmacokinetics and Pharmacodynamics of Disulfiram on Inducing Latent HIV-1 Transcription in a Phase IIb Trial. Clin Pharmacol Ther. 2019 Mar;105(3):692-702. doi: 10.1002/cpt.1220. Epub 2018 Oct 9. PMID 30137649
- [Background] Elliott JH, McMahon JH, Chang CC, Lee SA, Hartogensis W, Bumpus N, Savic R, Roney J, Hoh R, Solomon A, Piatak M, Gorelick RJ, Lifson J, Bacchetti P, Deeks SG, Lewin SR. Short-term administration of disulfiram for reversal of latent HIV infection: a phase 2 dose-escalation study. Lancet HIV. 2015 Dec;2(12):e520-9. doi: 10.1016/S2352-3018(15)00226-X. Epub 2015 Nov 17. PMID 26614966
- [Background] Jin Z, Du X, Xu Y, Deng Y, Liu M, Zhao Y, Zhang B, Li X, Zhang L, Peng C, Duan Y, Yu J, Wang L, Yang K, Liu F, Jiang R, Yang X, You T, Liu X, Yang X, Bai F, Liu H, Liu X, Guddat LW, Xu W, Xiao G, Qin C, Shi Z, Jiang H, Rao Z, Yang H. Structure of Mpro from SARS-CoV-2 and discovery of its inhibitors. Nature. 2020 Jun;582(7811):289-293. doi: 10.1038/s41586-020-2223-y. Epub 2020 Apr 9. PMID 32272481
- [Background] Lin MH, Moses DC, Hsieh CH, Cheng SC, Chen YH, Sun CY, Chou CY. Disulfiram can inhibit MERS and SARS coronavirus papain-like proteases via different modes. Antiviral Res. 2018 Feb;150:155-163. doi: 10.1016/j.antiviral.2017.12.015. Epub 2017 Dec 28. PMID 29289665
- [Background] Hu JJ, Liu X, Xia S, Zhang Z, Zhang Y, Zhao J, Ruan J, Luo X, Lou X, Bai Y, Wang J, Hollingsworth LR, Magupalli VG, Zhao L, Luo HR, Kim J, Lieberman J, Wu H. FDA-approved disulfiram inhibits pyroptosis by blocking gasdermin D pore formation. Nat Immunol. 2020 Jul;21(7):736-745. doi: 10.1038/s41590-020-0669-6. Epub 2020 May 4. PMID 32367036
- [Background] Lobo-Galo N, Terrazas-Lopez M, Martinez-Martinez A, Diaz-Sanchez AG. FDA-approved thiol-reacting drugs that potentially bind into the SARS-CoV-2 main protease, essential for viral replication. J Biomol Struct Dyn. 2021 Jun;39(9):3419-3427. doi: 10.1080/07391102.2020.1764393. Epub 2020 May 14. PMID 32364011
- [Derived] Saifi MA, Shaikh AS, Kaki VR, Godugu C. Disulfiram prevents collagen crosslinking and inhibits renal fibrosis by inhibiting lysyl oxidase enzymes. J Cell Physiol. 2022 May;237(5):2516-2527. doi: 10.1002/jcp.30717. Epub 2022 Mar 13. PMID 35285015

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Disulfiram 1000 mg: Participants in Cohort 1 receiving disulfiram will take 2 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
- Cohort 1: Placebo: This study will provide placebo comparator for disulfiram. Participants in Cohort 1 receiving placebo will take 2 capsules of placebo (each capsule contains only microcrystalline cellulose powder) per day for a total of 5 consecutive days.
- Cohort 2: Disulfiram 2000 mg: Participants in Cohort 2 receiving placebo will take 4 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
- Cohort 2: Placebo: Participants in Cohort 2 receiving placebo will take 4 capsules of placebo (each capsule contains only microcrystalline cellulose powder) per day for a total of 5 consecutive days.
Period: Overall Study
Arm/Group | Cohort 1 - Disulfiram 1000 mg | Cohort 1: Placebo | Cohort 2: Disulfiram 2000 mg | Cohort 2: Placebo
Started | 7 | 4 | 0 | 0
Completed | 7 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The trial stopped early so we were unable to enroll for Cohort 2.
Groups:
- Cohort 1: Disulfiram 1000 mg: This study will provide disulfiram. Participants in Cohort 1 receiving disulfiram will take 2 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Disulfiram 1000 mg | Cohort 1: Placebo | Cohort 2: Disulfiram 2000 mg | Cohort 2: Placebo | Total
Number analyzed (Participants) | 7 | 4 | 0 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 0 | 0 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12.5) | 43.5 (8) |  |  | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 |  |  | 7
  Male | 2 | 2 |  |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 |  |  | 4
  Not Hispanic or Latino | 4 | 3 |  |  | 7
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 1 | 0 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 1 | 0 |  |  | 1
  White | 5 | 4 |  |  | 9
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 |  |  | 11
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.6 (5.5) | 33.3 (2.2) |  |  | 28.4 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Impact of 5 Days of Disulfiram, as Measured by the Fold-change in Plasma Levels of Pro-inflammatory Cytokines (e.g, Interleukin 6, Interleukin 1-beta, Etc.).
Description: Change in plasma inflammatory biomarker levels (e.g., IL-6, IL-1b) at days 5, 15, and 31.
Time Frame: Day 0 and Day 31
Population: The trial stopped early so we were unable to enroll for Cohort 2.
Measure: Median (Inter-Quartile Range); unit: fold change
Groups:
- Cohort 1: Disulfiram 100 mg: This study will provide disulfiram. Participants in Cohort 1 receiving disulfiram will take 2 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
Arm/Group | Cohort 1: Disulfiram 100 mg | Cohort 1: Placebo | Cohort 2: Disulfiram 2000 mg | Cohort 2: Placebo
Number analyzed (Participants) | 7 | 4 | 0 | 0
fold change
  Change in IL-6 (pg/mL) Day 0 to 31 | -0.1186 [-0.2012 to -0.0246] | -0.0215 [-0.1202 to -0.0178] |  |
  Change in IL-1B (pg/mL) Day 0 to 31 | -0.1402 [-0.2583 to 0.0648] | 0.0268 [-0.0438 to 0.0399] |  |

2. Secondary Outcome: Virologic Impact of 5 Days of Disulfiram, as Measured by the Change in Copies of SARS-CoV-2 Virus Per mL Between Baseline and Day 31.
Description: Change in copies of SARS-CoV-2 PCR virus per mL between Baseline and Day 31.
Time Frame: Day 0 and Day 31
Population: The trial stopped early so we were unable to enroll for Cohort 2.
Measure: Mean (Standard Deviation); unit: copies/mL
Groups:
- Cohort 2: Disulfiram 2000 mg: Participants in Cohort 2 receiving disulfiram will take 4 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
Arm/Group | Cohort 1: Disulfiram 1000 mg | Cohort 1: Placebo | Cohort 2: Disulfiram 2000 mg | Cohort 2: Placebo
Number analyzed (Participants) | 7 | 4 | 0 | 0
copies/mL | -20.89 (9.84) | -20 (13.53) |  |

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: The safety and tolerability of a 5 day course of disulfiram. The number of adverse events and their grade will be determined for each participant.
Time Frame: Day 0 and Day 31
Population: The trial stopped early so we were unable to enroll for Cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Disulfiram 1000 mg | Cohort 1: Placebo | Cohort 2: Disulfiram 2000 mg | Cohort 2: Placebo
Number analyzed (Participants) | 7 | 4 | 0 | 0
Participants
  AE Grade 3 or Higher | 0 | 1 |  |
  AE Grade 1 or 2 | 4 | 1 |  |

4. Secondary Outcome: Change in COVID-19 Symptom Severity Score as Assessed by a 5-point Adapted Somatic Symptom Severity Score (SSS-8)
Description: The severity of COVID-19 symptoms will be recorded on a 5-point symptom severity scale at each visit for each participant. A question about how much the symptoms bother the participants will be asked. The participant will rank 1 as "not at all," 2 as "a little bit," 3 as "somewhat," 4 as "quite a bit" and 5 as "very much." Higher values represent worse outcomes. Scales are combined to compute a total score at Day 0 and Day 31. A change of the median is reported.
Time Frame: Day 0 and Day 31
Population: The trial stopped early so we were unable to enroll for Cohort 2.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Cohort 1: Disulfiram: This study will provide disulfiram. Participants in Cohort 1 receiving disulfiram will take 2 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
- Cohort 2: Disulfiram: Participants in Cohort 2 receiving placebo will take 4 capsules of disulfiram (each capsule contains 500 mg DSF plus 27.75 mg microcrystalline cellulose powder) per day for a total of 5 consecutive days.
Arm/Group | Cohort 1: Disulfiram | Cohort 1: Placebo | Cohort 2: Disulfiram | Cohort 2: Placebo
Number analyzed (Participants) | 7 | 4 | 0 | 0
units on a scale | -2.60 [-3.00 to 0.35] | -2.14 [-3.37 to -0.59] |  |

ADVERSE EVENTS:
Time Frame: The total duration of the study was approximately 6 months from August 18, 2021 to February 28, 2022. Each participant was assessed for 31 days during the duration of their enrollment in the study. There was one serious adverse event that lasted 5 days from September 6, 2021 to September 11, 2021.
Description: Systematic assessment through detailed questionnaires and principal investigator physical exam assessment was conducted at each visit.
Arm/Group | Cohort 1: Disulfiram | Cohort 1: Placebo | Cohort 2: Disulfiram | Cohort 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/7 | 1/4 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Disulfiram (N=7) | Cohort 1: Placebo (N=4) | Cohort 2: Disulfiram (N=0) | Cohort 2: Placebo (N=0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA | NA — Chest pain resulted in hospitalization for 5 days; no relationship to study drug and was resolved
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Disulfiram (N=7) | Cohort 1: Placebo (N=4) | Cohort 2: Disulfiram (N=0) | Cohort 2: Placebo (N=0)
Dehydration (Renal and urinary disorders) | 1 (1) | 0 (0) | NA | NA — dehydration for 1 day; not related to study drug and was resolved
Black stool and post viral cough syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA | NA — Mild severity of black stool and not related to study drug Moderate severity of post viral cough syndrome and not related to study drug
GI (nausea/vomiting), fever, chills, congestion, sore throat, back pain, muscle ache, headache (General disorders) | 1 (1) | 0 (0) | NA | NA — All symptoms were mild severity and not related to study drug
Smell and taste (General disorders) | 1 (1) | 0 (0) | NA | NA — Mild severity lasting 11 days until resolved; not related to study drug
Smell/taste, gas, back pain (General disorders) | 1 (1) | 0 (0) | NA | NA — All mild severity; not related to study drug Back pain lasted 1 day until resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT04485130/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT04485130/ICF_001.pdf